CLINICAL TRIAL: NCT04592419
Title: A Prospective, Randomized, Double-masked, Active Comparator-controlled, Multi-center, Two-arm, Phase 3 Study to Evaluate the Efficacy and Safety of Intravitreal KSI-301 Compared With Intravitreal Aflibercept in Participants With Visual Impairment Due to Treatment-naïve Macular Edema Secondary to Retinal Vein Occlusion (RVO)
Brief Title: A Study to Evaluate the Efficacy, Durability, and Safety of KSI-301 Compared to Aflibercept in Patients With Macular Edema Due to Retinal Vein Occlusion (RVO)
Acronym: BEACON
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kodiak Sciences Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KS301P103; 2020-001061-37 (EudraCT Number)
Record Dates: First submitted 2020-10-12; First posted 2020-10-19 (Actual); Results first posted 2024-06-06 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Macular Edema; Retinal Vein Occlusion
Keywords: RVO; Kodiak; KSI-301; Vascular endothelial growth factor; Anti-VEGF; VEGF; Antibody biopolymer conjugate; Retinal Degeneration; Retinal Diseases; Eye Diseases; Vision Disorders; Vision, low; Aflibercept; Eylea
MeSH Terms: conditions — Macular Edema; Retinal Vein Occlusion; Retinal Degeneration; Retinal Diseases; Eye Diseases; Vision Disorders; Vision, Low | interventions — aflibercept

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 1:1 into one of two treatment arms: KSI-301 or aflibercept.
  Participants in the Extension Phase will be treated with KSI-301.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: For masking purposes, sham injections will be administered at every monthly visit if an active treatment is not administered. To preserve masking, two investigators are required for this study. The masked Investigator will be responsible for the examinations and safety assessments. The unmasked Investigator will perform the injections and post-treatment assessments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- KSI-301 (Arm A) (Experimental): Intravitreal injection of KSI-301 (5 mg) at Day 1, Week 4, and once every 8 weeks through Week 20 followed by an individualized dosing regimen of Intravitreal injection of KSI-301 (5 mg) from Week 24 to Week 44.
  In the Extension Phase, participants randomized to KSI-301 (5 mg) in the Primary Study will continue to receive KSI-301 (5 mg) based on protocol-defined disease activity criteria.
  Interventions: Drug: KSI-301; Other: Sham Procedure
- Aflibercept (Arm B) (Active Comparator): Intravitreal injection of aflibercept (2 mg) once every 4 through Week 20 followed by an individualized dosing regimen of Intravitreal injection of Aflibercept (2 mg) once every 4 weeks from Week 24 to Week 44.
  In the Extension Phase, participants randomized to aflibercept in the Primary Study will cross over to treatment with KSI-301 (5 mg). They will receive their first dose of KSI-301 (5 mg) at Week 48 and will receive additional treatment with KSI-301 (5 mg) based on protocol-defined disease activity criteria.
  Interventions: Drug: Aflibercept; Other: Sham Procedure

INTERVENTIONS:
Drug: KSI-301 — Intravitreal Injection
  Arms: KSI-301 (Arm A)
Drug: Aflibercept — Intravitreal Injection
  Other Names: Eylea
  Arms: Aflibercept (Arm B)
Other: Sham Procedure — The sham is a procedure that mimics an intravitreal injection. It involves pressing the blunt end of an empty syringe (without a needle) against the anesthetized eye. It will be administered to participants in both treatments arms at applicable visits to maintain masking.

SUMMARY:
This Phase 3 study will evaluate the efficacy, durability, and safety of KSI-301 compared to aflibercept, in participants with macular edema due to treatment-naïve branch (BRVO) or central retinal vein occlusion (CRVO).

DETAILED DESCRIPTION:
This is a Phase 3, prospective, randomized, double-masked, two-arm, multi-center non-inferiority study evaluating the efficacy and safety of repeated intravitreal dosing of KSI-301 5 mg in participants with visual impairment due to treatment-naïve macular edema secondary to RVO (either branch or central type).

The primary endpoint will be assessed at Week 24; additional secondary endpoints for efficacy will be assessed at Week 24 and Week 48.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent prior to participation in the study.
2. Treatment-naïve macular edema of 6 months duration or less due to CRVO or BRVO. Participants with hemiretinal vein occlusion will be included as CRVO.
3. BCVA ETDRS letter score between 80 and 25 (20/25 to 20/320 Snellen equivalent), inclusive in the Study Eye.
4. CST of ≥ 320 microns on SD-OCT (Heidelberg Spectralis or equivalent on other OCT instruments) as determined by the Reading Center
5. Decrease in vision determined by the Investigator to be primarily the result of ME secondary to RVO.
6. Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

1. Macular edema in the Study Eye for reasons other than RVO
2. Active iris or angle neovascularization, neovascular glaucoma, neovascularization of the optic disc, retinal neovascularization or vitreous hemorrhage in the Study Eye.
3. Uncontrolled glaucoma in the Study Eye.
4. Active retinal disease other than the condition under investigation in the Study Eye.
5. Any history or evidence of a concurrent ocular condition present, that in the opinion of the Investigator could require either medical or surgical intervention alter visual acuity during the study
6. Active or suspected ocular or periocular infection or inflammation
7. Any prior use of an approved or investigational treatment for macular edema secondary to RVO in the Study Eye (e.g. anti-VEGF, intraocular or periocular steroids, macular laser photocoagulation).
8. Women who are pregnant or lactating or intending to become pregnant during the study.
9. Uncontrolled blood pressure defined as a systolic value ≥ 180 mmHg or diastolic value ≥100 mmHg while at rest
10. Recent history (within the 6 months prior to screening) of myocardial infarction, stroke, transient ischemic attack, acute congestive heart failure or any acute coronary event.
11. History of a medical condition that, in the judgment of the Investigator, would preclude scheduled study visits, completion of the study, or a safe administration of investigational product.
12. Other protocol-specified exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 568 (Actual)
Dates: Start 2020-09-25 (Actual); Primary Completion 2022-06-10 (Actual); Study Completion 2023-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Velazquez-Martin, MD, Study Director — Kodiak Sciences Inc
Locations (141):
- United States (81):
  - Northwest Arkansas Retina Associates, Phoenix, Arizona
  - Retinal Research Institute, LLC, Phoenix, Arizona
  - Retina Vitreous Associates, Beverly Hills, California
  - Eye Medical Center of Fresno, Fresno, California
  - Retina Consultants of Orange County, Fullerton, California
  - UCSD Jacobs Retina Center, La Jolla, California
  - Northern California Retina Vitreous Associates, Mountain View, California
  - Retina Consultants of San Diego, Poway, California
  - Retina Consultants of Southern California, Redlands, California
  - Retinal Consultants Medical Group Inc, Sacramento, California
  - Orange County Retina Medical Group, Santa Ana, California
  - California Retina Consultants, Santa Maria, California
  - Colorado Retina Associates PC, Lakewood, Colorado
  - Conneticut Eye Consultants, Danbury, Connecticut
  - Retina Group of New England, Waterford, Connecticut
  - Florida Eye Clinic, Altamonte Springs, Florida
  - Retina Group of Florida, Boca Raton, Florida
  - Florida Eye Microsurgical Institute, Boynton Beach, Florida
  - The Macula Center/ Blue Ocean Clinical Research, Clearwater, Florida
  - Rand Eye Institute, Deerfield Beach, Florida
  - National Ophthalmic Research Institute, Fort Myers, Florida
  - Vitreo Retinal Associates, Gainesville, Florida
  - Florida Eye Associates, Melbourne, Florida
  - Florida Retina Institute, Orlando, Florida
  - Retina Specialty Institute, Pensacola, Florida
  - Fort Lauderdale Eye Institute, Plantation, Florida
  - Southern Vitreoretinal Associates, Tallahassee, Florida
  - Retina Associates of Florida, Tampa, Florida
  - Center for Retina & Macular Disease, Winter Haven, Florida
  - Southeast Retina Center, Augusta, Georgia
  - Springfield Clinic LLP, Springfield, Illinois
  - Talley Eye, Evansville, Indiana
  - Wolfe Eye Clinic, West Des Moines, Iowa
  - Retina Associates PA, Lenexa, Kansas
  - Vitreo Retinal Consultants and Surgeons, Wichita, Kansas
  - Retina Associates of Kentucky, Lexington, Kentucky
  - Maine Eye Center, Portland, Maine
  - Retina Group of Washington, Chevy Chase, Maryland
  - Cumberland Valley Retina Consultants PC, Hagerstown, Maryland
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Vitreo Retinal Associates PC, Worcester, Massachusetts
  - Foundation for Vision Research, Grand Rapids, Michigan
  - Associated Retinal Consultants PC, Royal Oak, Michigan
  - Vitreoretinal Surgery PA, Edina, Minnesota
  - Retina Consultants of NV, Henderson, Nevada
  - Sierra Eye Associates, Reno, Nevada
  - The Retina Center of New Jersey, Bloomfield, New Jersey
  - NJ Retina, Teaneck, New Jersey
  - Vitreo Retinal Consultants, Hauppauge, New York
  - Retina-Vitreous Surgeons of Central NY, Liverpool, New York
  - Ocli Vision, Oceanside, New York
  - Retina Associates of Western NY, Rochester, New York
  - Asheville Eye Associates, Asheville, North Carolina
  - Charlotte Eye Ear Nose & Throat Associates, P.A., Charlotte, North Carolina
  - Retina Associates of Cleveland, Beachwood, Ohio
  - Retina Associates of Cleveland, Cleveland, Ohio
  - Retina Northwest, Portland, Oregon
  - Retina Consultants, LLC, Salem, Oregon
  - Cascade Medical Research Institute, Springfield, Oregon
  - Retina Research of Beaufort, Beaufort, South Carolina
  - Retina Consultants of Carolina, Greenville, South Carolina
  - Charleston Neuroscience Institute, Ladson, South Carolina
  - Pametto Retina Center, West Columbia, South Carolina
  - Black Hills Regional Eye Institute, Rapid City, South Dakota
  - Charles Retina Institute, Germantown, Tennessee
  - Southeastern Retina Associates PC, Knoxville, Tennessee
  - Tennessee Retina PC, Nashville, Tennessee
  - Retina Research Institute of Texas, Abilene, Texas
  - Austin Research Center for Retina, Austin, Texas
  - Austin Retina Associates, Austin, Texas
  - Retina Research Center, Austin, Texas
  - Retina Consultants of Texas, Houston, Texas
  - Retina Consultants of Texas - (Katy), Katy, Texas
  - Texas Retina Associates, Plano, Texas
  - Austin Retina Associates (Round Rock), Round Rock, Texas
  - Medical Center Ophthalmology Associates, San Antonio, Texas
  - Retina Consultants of Texas - (Woodlands), The Woodlands, Texas
  - Strategic Clinical Research Group, LLC, Willow Park, Texas
  - Retina Institute of Virginia, Richmond, Virginia
  - Retina Center Northwest, Silverdale, Washington
  - Spokane Eye, Spokane, Washington
- Czechia (3):
  - OFTEX s.r.o., Pardubice
  - Vseobecna Fakultni, Prague
  - Lekarna BENU, Prague
- France (8):
  - CHRU Dijon Complexe Du Bocage, Dijon, Côte-d'Or
  - Centre Hospitalier Universitaire de Bordeaux, Hopital Pellegrin, Bordeaux, Gironde
  - Hôpital de La Croix Rousse, Lyon, Rhône
  - Centre Hospitalier Intercommunal de Créteil, Créteil
  - Centre Paradis Monticelli, Marseille
  - Hôpital Lariboisière - Service Pharmacie, Paris
  - Fondation Rothschild, Paris
  - CHRU de Poitiers La Miletrie, Poitiers
- Germany (4):
  - Universitätsklinikum Regensburg, Regensburg, Bavaria
  - Dietrich Bonhoeffer Klinikum Neubrandenburg, Neubrandenburg, Mecklenburg-Vorpommern
  - St. Elisabeth Krankenhaus, Cologne, North Rhine-Westphalia
  - Miriam Kannenbaeumer or Andrea Koschinski, Münster, North Rhine-Westphalia
- Hungary (5):
  - MH EK Honvedkorhaz SzemEszeti Osztaly, Budapest
  - Semmelweis Egyetem, Budapest
  - Bajcsy-Zsilinszky Korhaz es Rendelointezet, Budapest
  - Budapest Retina Associates Kft, Budapest
  - Jahn Ferenc Dél-Pesti Kórház és Rendelointézet, Budapest
- Israel (9):
  - Bnai Zion, Haifa
  - Rambam MC, Haifa
  - Hadassah University Hospital, Jerusalem
  - Meir MC, Kfar Saba
  - Rabin Medical Center, Petah Tikva
  - Kaplan MC, Rehovot
  - Tel Aviv Sourasky Medical Center, Tel Aviv
  - Assuta HaShalom, Tel Aviv
  - Shamir Medical Center Assaf Harofeh, Tzrifin
- Italy (5):
  - Ospedale Clinicizzato SS Annunziata, Chieti, Abruzzo
  - Fondazione PTV Policlinico Tor Vergata, Rome, Lazio
  - Fondazione Policlinico Universitario A Gemelli, Rome, Lazio
  - Ospedale San Raffaele S.r.l. - PPDS, Milan, Lombardy
  - Azienda Sanitaria Universitaria Integrata di Udine - PO Universitario Santa Maria della Misericordia, Udine
- Latvia (4):
  - Signes Ozolinas Doctor Praxis In Ophthalmology, Jelgava
  - Pauls Stradins Clinical University Hospital, Riga
  - Riga Eastern Clinical University Hospital Clinic Bikernieki, Riga
  - Latvian American Eye Center, Riga
- Poland (6):
  - Optimum Profesorskie Centrum Okulistyki, Gdansk, Pomeranian Voivodeship
  - Uniwersyteckie Centrum Kliniczne Im. Prof. K. Gibinskiego Slaskiego Uniwersytetu Medycznego w Katowi, Katowice, Silesian Voivodeship
  - Gabinet Okulistyczny Prof. Edward Wylegala, Katowice, Silesian Voivodeship
  - Oftalmika Sp. z o.o., Bydgoszcz
  - Dr Nowosielska Okulistyka i Chirurgia Oka, Warsaw
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza Radeckiego we Wroclawiu, Wroclaw
- Emanuelli Research & Development Center LLC, Arecibo, Puerto Rico
- Slovakia (5):
  - Fakultna nemocnica s poliklinikou F. D. Roosevelta, Banská Bystrica
  - Univerzitna nemocnica Bratislava, Bratislava
  - Uvea Klinika, S.R.O., Martin
  - Nemocnica s poliklinikou Trebisov a.s., Trebišov
  - Fakultna nemocnica Trencin, Trencín
- Spain (10):
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitari General de Catalunya - Grupo Quironsalud, Sant Cugat del Vallès, Barcelona
  - Hospital Universitario Puerta de Hierro - Majadahonda, Majadahonda, Madrid
  - Hospital dos de Maig, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Instituto Clinico Quirurgico de Oftalmologia, Bilbao
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
  - Hospital Universitario Rio Hortega, Valladolid
  - Hospital Clinico Universitario Lozano Blesa, Zaragoza
  - Hospital Universitario Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on physician referral at 138 medical centers between September 2020 and December 2021. The first participant was enrolled on 25 September 2020 and the last on 15 December 2021.
Pre-assignment Details: Of 752 enrolled participants, 568 met eligibility criteria and were randomized to treatment.
Groups:
- KSI-301 (Arm A): Intravitreal injection of KSI-301 (5 mg) at Day 1, Week 4, and once every 8 weeks through Week 20 followed by an individualized dosing regimen of Intravitreal injection of KSI-301 (5 mg) from Week 24 to Week 44.
  In the Extension Phase, participants randomized to KSI-301 (5 mg) in the Primary Study will continue to receive KSI-301 (5 mg) based on protocol-defined disease activity criteria.
  KSI-301: Intravitreal Injection
  Sham Procedure: The sham is a procedure that mimics an intravitreal injection. It involves pressing the blunt end of an empty syringe (without a needle) against the anesthetized eye. It will be administered to participants in both treatments arms at applicable visits to maintain masking.
- Aflibercept (Arm B): Intravitreal injection of aflibercept (2 mg) once every 4 weeks through Week 20 followed by an individualized dosing regimen of Intravitreal injection of Aflibercept (2 mg) once every 4 weeks from Week 24 to Week 44.
  In the Extension Phase, participants randomized to aflibercept in the Primary Study will cross over to treatment with KSI-301 (5 mg). They will receive their first dose of KSI-301 (5 mg) at Week 48 and will receive additional treatment with KSI-301 (5 mg) based on protocol-defined disease activity criteria.
  Aflibercept: Intravitreal Injection
  Sham Procedure: The sham is a procedure that mimics an intravitreal injection. It involves pressing the blunt end of an empty syringe (without a needle) against the anesthetized eye. It will be administered to participants in both treatments arms at applicable visits to maintain masking.
Period: Primary Study (Through Year 1)
Arm/Group | KSI-301 (Arm A) | Aflibercept (Arm B)
Started | 284 | 284
Completed Treatment at Week 20 | 270 | 274
Did Not Discontinue Treatment Before Week 24 | 270 | 276
Did Not Discontinue Study Before Week 24 | 275 | 276
Completed | 255 (Completed is defined as those who completed through Week 48.) | 255 (Completed is defined as those who completed through Week 48.)
Not Completed | 29 | 29
Not completed — Adverse Event | 10 | 3
Not completed — Non-compliance with Study Schedule | 0 | 1
Not completed — Withdrawal by Subject | 7 | 13
Not completed — Lost to Follow-up | 5 | 5
Not completed — Progressive Disease | 1 | 1
Not completed — Sponsor Request | 4 | 5
Not completed — Participant left the country | 2 | 0
Not completed — Participant moved to another city with no available site | 0 | 1
Period: Open-Label Extension Period
Arm/Group | KSI-301 (Arm A) | Aflibercept (Arm B)
Started | 216 | 228
Completed | 135 | 130
Not Completed | 81 | 98
Not completed — Adverse Event | 1 | 2
Not completed — Non-compliance with Study Schedule | 1 | 0
Not completed — Withdrawal by Subject | 5 | 7
Not completed — Lost to Follow-up | 1 | 5
Not completed — Sponsor Request | 73 | 84

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (Week 24 or 48) includes all randomized participants who received at least one treatment injection in the first 24/48 weeks and using all available post baseline measurements up to Week 24/48 or until the participant discontinues study treatment. Number analyzed by visit is equal to the number of participants who had data available at that respective visit.
Groups:
- Aflibercept (Arm B): Intravitreal injection of aflibercept (2 mg) once every 4 through Week 20 followed by an individualized dosing regimen of Intravitreal injection of Aflibercept (2 mg) once every 4 weeks from Week 24 to Week 44.
  In the Extension Phase, participants randomized to aflibercept in the Primary Study will cross over to treatment with KSI-301 (5 mg). They will receive their first dose of KSI-301 (5 mg) at Week 48 and will receive additional treatment with KSI-301 (5 mg) based on protocol-defined disease activity criteria.
  Aflibercept: Intravitreal Injection
  Sham Procedure: The sham is a procedure that mimics an intravitreal injection. It involves pressing the blunt end of an empty syringe (without a needle) against the anesthetized eye. It will be administered to participants in both treatments arms at applicable visits to maintain masking.
- Total: Total of all reporting groups
Arm/Group | KSI-301 (Arm A) | Aflibercept (Arm B) | Total
Number analyzed (Participants) | 284 | 284 | 568
Age, Customized [Count of Participants; unit: Participants]
  18-64 years | 126 | 142 | 268
  65-74 years | 94 | 86 | 180
  75-84 years | 50 | 41 | 91
  ≥ 85 years | 14 | 15 | 29
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 141 | 138 | 279
  Male | 143 | 146 | 289
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 5 | 5 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 23 | 17 | 40
  White | 240 | 245 | 485
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 15 | 14 | 29
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 31 | 29 | 60
  Not Hispanic or Latino | 242 | 246 | 488
  Choose Not to Respond | 11 | 9 | 20
Geographic Region [Count of Participants; unit: Participants]
  North America | 193 | 193 | 386
  Rest of World | 91 | 91 | 182
Blood Pressure at Baseline [Mean (Standard Deviation); unit: mmHG]
  Systolic | 139.1 (16.66) | 138.7 (16.42) | 138.9 (16.52)
  Diastolic | 82.8 (8.71) | 82.6 (9.33) | 82.7 (9.02)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Best Corrected Visual Acuity (BCVA) From Day 1 to Week 24 in BRVO Participants.
Description: BCVA as a continuous variable measured at each study visit using the Early Treatment Diabetic Retinopathy Study (ETDRS) BCVA approach.
Time Frame: Day 1 to Week 24
Population: Full Analysis Set (Week 24) includes all randomized participants who received at least one treatment injection in the first 24 weeks and using all available post baseline measurements up to Week 24 or until the participant discontinues study treatment.
Measure: Least Squares Mean (Standard Error); unit: ETDRS Letters
Arm/Group | KSI-301 (Arm A) | Aflibercept (Arm B)
Number analyzed (Participants) | 220 | 218
ETDRS Letters | 14.2 (.81) | 15.6 (.79)
Statistical Analysis 1: Comparison: KSI-301 (Arm A) vs Aflibercept (Arm B); Test type: Non-Inferiority — The maximum clinically acceptable true difference between KSI-301 and aflibercept among BRVO participants to be considered non-inferior is 4.5 ETDRS letters, i.e. the non-inferiority margin (NI) is 4.5 letters; p = .0004, Mixed Models Analysis; MMRM model with treatment, visit, treatment × visit interaction, baseline BCVA, disease duration, and geographical location as covariates; Adjusted mean difference = -1.4, 95.02% CI 2-sided [-3.11 to 0.30], Standard Error of Mean .87

2. Primary Outcome: Mean Change in Best Corrected Visual Acuity (BCVA) From Day 1 to Week 24 in All RVO Patients.
Description: as for outcome 1
Time Frame: Day 1 to Week 24
Population: Full Analysis Set (Week 24) includes all randomized subjects who received at least one treatment injection in the first 24 weeks and using all available post baseline measurements up to Week 24 or until the subject discontinues study treatment.
Measure: Least Squares Mean (Standard Error); unit: ETDRS Letters
Arm/Group | KSI-301 (Arm A) | Aflibercept (Arm B)
Number analyzed (Participants) | 284 | 284
ETDRS Letters | 13.0 (.83) | 15.5 (.81)
Statistical Analysis 1: Comparison: KSI-301 (Arm A) vs Aflibercept (Arm B); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = .0243, Mixed Models Analysis; MMRM model treatment, visit, treatment × visit interaction, RVO subtype, baseline BCVA, disease duration, and geographical location as covariates; Adjusted mean difference = -2.5, 95.02% CI 2-sided [-4.24 to -0.71], Standard Error of Mean .90

3. Secondary Outcome: Mean Change From Baseline in BCVA (ETDRS Letters) by Visit Over Time up to Week 48 for All RVO Participants.
Description: as for outcome 1
Time Frame: Day 1 - Week 48
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: ETDRS Letters
Arm/Group | KSI-301 (Arm A) | Aflibercept (Arm B)
Number analyzed (Participants) | 284 | 284
ETDRS Letters
  Week 1: number analyzed (Participants) | 280 | 275
  Week 1 | 7.7 (9.25) | 7.9 (7.74)
  Week 4: number analyzed (Participants) | 279 | 275
  Week 4 | 8.9 (9.89) | 11.2 (10.01)
  Week 8: number analyzed (Participants) | 273 | 278
  Week 8 | 11.4 (10.38) | 13.5 (9.78)
  Week 12: number analyzed (Participants) | 276 | 277
  Week 12 | 10.0 (12.58) | 14.2 (10.05)
  Week 16: number analyzed (Participants) | 270 | 272
  Week 16 | 12.7 (11.99) | 14.9 (10.52)
  Week 20: number analyzed (Participants) | 263 | 269
  Week 20 | 12.4 (12.29) | 15.3 (11.86)
  Week 24: number analyzed (Participants) | 261 | 267
  Week 24 | 14.0 (11.42) | 15.6 (11.54)
  Week 28: number analyzed (Participants) | 257 | 264
  Week 28 | 12.8 (11.85) | 14.1 (12.90)
  Week 32: number analyzed (Participants) | 250 | 257
  Week 32 | 13.3 (11.55) | 13.8 (12.46)
  Week 36: number analyzed (Participants) | 252 | 259
  Week 36 | 13.1 (11.52) | 13.5 (11.96)
  Week 40: number analyzed (Participants) | 252 | 257
  Week 40 | 13.9 (11.51) | 13.9 (12.87)
  Week 44: number analyzed (Participants) | 244 | 256
  Week 44 | 13.6 (11.26) | 13.7 (13.11)
  Week 48: number analyzed (Participants) | 247 | 252
  Week 48 | 13.5 (12.10) | 14.2 (13.64)

4. Secondary Outcome: Percentage of Participants Who Gain ≥ 5, ≥10 and ≥15 Letters From Baseline Over Time up to Week 48 for All RVO Participants.
Description: Number of participants in each treatment arm who meet specified criteria at each visit from Week 1 through Week 48. Percentages are 100*n/N.
Time Frame: Day 1 - Week 48
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | KSI-301 (Arm A) | Aflibercept (Arm B)
Number analyzed (Participants) | 284 | 284
Participants
  Participants who gain ≥ 5 letters from baseline to Week 1.: number analyzed (Participants) | 280 | 275
  Participants who gain ≥ 5 letters from baseline to Week 1. | 176 | 176
  Participants who gain ≥ 5 letters from baseline to Week 4.: number analyzed (Participants) | 279 | 275
  Participants who gain ≥ 5 letters from baseline to Week 4. | 197 | 202
  Participants who gain ≥ 5 letters from baseline to Week 8.: number analyzed (Participants) | 273 | 278
  Participants who gain ≥ 5 letters from baseline to Week 8. | 211 | 233
  Participants who gain ≥ 5 letters from baseline to Week 12.: number analyzed (Participants) | 276 | 277
  Participants who gain ≥ 5 letters from baseline to Week 12. | 198 | 237
  Participants who gain ≥ 5 letters from baseline to Week 16.: number analyzed (Participants) | 270 | 272
  Participants who gain ≥ 5 letters from baseline to Week 16. | 222 | 240
  Participants who gain ≥ 5 letters from baseline to Week 20.: number analyzed (Participants) | 263 | 269
  Participants who gain ≥ 5 letters from baseline to Week 20. | 199 | 235
  Participants who gain ≥ 5 letters from baseline to Week 24.: number analyzed (Participants) | 261 | 267
  Participants who gain ≥ 5 letters from baseline to Week 24. | 215 | 233
  Participants who gain ≥ 5 letters from baseline to Week 28.: number analyzed (Participants) | 257 | 264
  Participants who gain ≥ 5 letters from baseline to Week 28. | 206 | 211
  Participants who gain ≥ 5 letters from baseline to Week 32.: number analyzed (Participants) | 250 | 257
  Participants who gain ≥ 5 letters from baseline to Week 32. | 200 | 213
  Participants who gain ≥ 5 letters from baseline to Week 36.: number analyzed (Participants) | 252 | 259
  Participants who gain ≥ 5 letters from baseline to Week 36. | 205 | 212
  Participants who gain ≥ 5 letters from baseline to Week 40.: number analyzed (Participants) | 252 | 257
  Participants who gain ≥ 5 letters from baseline to Week 40. | 210 | 215
  Participants who gain ≥ 5 letters from baseline to Week 44.: number analyzed (Participants) | 244 | 256
  Participants who gain ≥ 5 letters from baseline to Week 44. | 196 | 211
  Participants who gain ≥ 5 letters from baseline to Week 48.: number analyzed (Participants) | 247 | 252
  Participants who gain ≥ 5 letters from baseline to Week 48. | 199 | 206
  Participants who gain ≥ 10 letters from baseline to Week 1.: number analyzed (Participants) | 280 | 275
  Participants who gain ≥ 10 letters from baseline to Week 1. | 94 | 91
  Participants who gain ≥ 10 letters from baseline to Week 4.: number analyzed (Participants) | 279 | 275
  Participants who gain ≥ 10 letters from baseline to Week 4. | 120 | 145
  Participants who gain ≥ 10 letters from baseline to Week 8.: number analyzed (Participants) | 273 | 278
  Participants who gain ≥ 10 letters from baseline to Week 8. | 151 | 175
  Participants who gain ≥ 10 letters from baseline to Week 12.: number analyzed (Participants) | 276 | 277
  Participants who gain ≥ 10 letters from baseline to Week 12. | 141 | 179
  Participants who gain ≥ 10 letters from baseline to Week 16.: number analyzed (Participants) | 270 | 272
  Participants who gain ≥ 10 letters from baseline to Week 16. | 168 | 181
  Participants who gain ≥ 10 letters from baseline to Week 20.: number analyzed (Participants) | 263 | 269
  Participants who gain ≥ 10 letters from baseline to Week 20. | 168 | 183
  Participants who gain ≥ 10 letters from baseline to Week 24.: number analyzed (Participants) | 261 | 267
  Participants who gain ≥ 10 letters from baseline to Week 24. | 177 | 188
  Participants who gain ≥ 10 letters from baseline to Week 28.: number analyzed (Participants) | 257 | 264
  Participants who gain ≥ 10 letters from baseline to Week 28. | 160 | 168
  Participants who gain ≥ 10 letters from baseline to Week 32.: number analyzed (Participants) | 250 | 257
  Participants who gain ≥ 10 letters from baseline to Week 32. | 164 | 172
  Participants who gain ≥ 10 letters from baseline to Week 36.: number analyzed (Participants) | 252 | 259
  Participants who gain ≥ 10 letters from baseline to Week 36. | 158 | 162
  Participants who gain ≥ 10 letters from baseline to Week 40.: number analyzed (Participants) | 252 | 257
  Participants who gain ≥ 10 letters from baseline to Week 40. | 167 | 162
  Participants who gain ≥ 10 letters from baseline to Week 44.: number analyzed (Participants) | 244 | 256
  Participants who gain ≥ 10 letters from baseline to Week 44. | 156 | 164
  Participants who gain ≥ 10 letters from baseline to Week 48.: number analyzed (Participants) | 247 | 252
  Participants who gain ≥ 10 letters from baseline to Week 48. | 159 | 164
  Participants who gain ≥ 15 letters from baseline to Week 1.: number analyzed (Participants) | 280 | 275
  Participants who gain ≥ 15 letters from baseline to Week 1. | 46 | 49
  Participants who gain ≥ 15 letters from baseline to Week 4.: number analyzed (Participants) | 279 | 275
  Participants who gain ≥ 15 letters from baseline to Week 4. | 69 | 85
  Participants who gain ≥ 15 letters from baseline to Week 8.: number analyzed (Participants) | 273 | 278
  Participants who gain ≥ 15 letters from baseline to Week 8. | 92 | 111
  Participants who gain ≥ 15 letters from baseline to Week 12.: number analyzed (Participants) | 276 | 277
  Participants who gain ≥ 15 letters from baseline to Week 12. | 83 | 119
  Participants who gain ≥ 15 letters from baseline to Week 16.: number analyzed (Participants) | 270 | 272
  Participants who gain ≥ 15 letters from baseline to Week 16. | 109 | 131
  Participants who gain ≥ 15 letters from baseline to Week 20.: number analyzed (Participants) | 263 | 269
  Participants who gain ≥ 15 letters from baseline to Week 20. | 109 | 137
  Participants who gain ≥ 15 letters from baseline to Week 24.: number analyzed (Participants) | 261 | 267
  Participants who gain ≥ 15 letters from baseline to Week 24. | 121 | 138
  Participants who gain ≥ 15 letters from baseline to Week 28.: number analyzed (Participants) | 257 | 264
  Participants who gain ≥ 15 letters from baseline to Week 28. | 111 | 118
  Participants who gain ≥ 15 letters from baseline to Week 32.: number analyzed (Participants) | 250 | 257
  Participants who gain ≥ 15 letters from baseline to Week 32. | 113 | 113
  Participants who gain ≥ 15 letters from baseline to Week 36.: number analyzed (Participants) | 252 | 259
  Participants who gain ≥ 15 letters from baseline to Week 36. | 108 | 112
  Participants who gain ≥ 15 letters from baseline to Week 40.: number analyzed (Participants) | 252 | 257
  Participants who gain ≥ 15 letters from baseline to Week 40. | 107 | 120
  Participants who gain ≥ 15 letters from baseline to Week 44.: number analyzed (Participants) | 244 | 256
  Participants who gain ≥ 15 letters from baseline to Week 44. | 111 | 116
  Participants who gain ≥ 15 letters from baseline to Week 48.: number analyzed (Participants) | 247 | 252
  Participants who gain ≥ 15 letters from baseline to Week 48. | 112 | 120

5. Secondary Outcome: Percentage of Participants Who Lose ≥ 5, ≥10 and ≥15 ETDRS Letters From Baseline Over Time up to Week 48 for All RVO Participants
Description: as for outcome 4
Time Frame: Day 1 - Week 48
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | KSI-301 (Arm A) | Aflibercept (Arm B)
Number analyzed (Participants) | 284 | 284
Participants
  Participants who lose ≥ 5 letters from baseline to Week 1.: number analyzed (Participants) | 280 | 275
  Participants who lose ≥ 5 letters from baseline to Week 1. | 5 | 6
  Participants who lose ≥ 5 letters from baseline to Week 4.: number analyzed (Participants) | 279 | 275
  Participants who lose ≥ 5 letters from baseline to Week 4. | 19 | 7
  Participants who lose ≥ 5 letters from baseline to Week 8.: number analyzed (Participants) | 273 | 278
  Participants who lose ≥ 5 letters from baseline to Week 8. | 14 | 3
  Participants who lose ≥ 5 letters from baseline to Week 12.: number analyzed (Participants) | 276 | 277
  Participants who lose ≥ 5 letters from baseline to Week 12. | 18 | 3
  Participants who lose ≥ 5 letters from baseline to Week 16.: number analyzed (Participants) | 270 | 272
  Participants who lose ≥ 5 letters from baseline to Week 16. | 13 | 5
  Participants who lose ≥ 5 letters from baseline to Week 20.: number analyzed (Participants) | 263 | 269
  Participants who lose ≥ 5 letters from baseline to Week 20. | 17 | 8
  Participants who lose ≥ 5 letters from baseline to Week 24.: number analyzed (Participants) | 261 | 267
  Participants who lose ≥ 5 letters from baseline to Week 24. | 13 | 7
  Participants who lose ≥ 5 letters from baseline to Week 28.: number analyzed (Participants) | 257 | 264
  Participants who lose ≥ 5 letters from baseline to Week 28. | 16 | 10
  Participants who lose ≥ 5 letters from baseline to Week 32.: number analyzed (Participants) | 250 | 257
  Participants who lose ≥ 5 letters from baseline to Week 32. | 14 | 9
  Participants who lose ≥ 5 letters from baseline to Week 36.: number analyzed (Participants) | 252 | 259
  Participants who lose ≥ 5 letters from baseline to Week 36. | 16 | 11
  Participants who lose ≥ 5 letters from baseline to Week 40.: number analyzed (Participants) | 252 | 257
  Participants who lose ≥ 5 letters from baseline to Week 40. | 13 | 14
  Participants who lose ≥ 5 letters from baseline to Week 44.: number analyzed (Participants) | 244 | 256
  Participants who lose ≥ 5 letters from baseline to Week 44. | 10 | 15
  Participants who lose ≥ 5 letters from baseline to Week 48.: number analyzed (Participants) | 247 | 252
  Participants who lose ≥ 5 letters from baseline to Week 48. | 18 | 15
  Participants who lose ≥ 10 letters from baseline to Week 1.: number analyzed (Participants) | 280 | 275
  Participants who lose ≥ 10 letters from baseline to Week 1. | 3 | 1
  Participants who lose ≥ 10 letters from baseline to Week 4.: number analyzed (Participants) | 279 | 275
  Participants who lose ≥ 10 letters from baseline to Week 4. | 4 | 1
  Participants who lose ≥ 10 letters from baseline to Week 8.: number analyzed (Participants) | 273 | 278
  Participants who lose ≥ 10 letters from baseline to Week 8. | 6 | 1
  Participants who lose ≥ 10 letters from baseline to Week 12.: number analyzed (Participants) | 276 | 277
  Participants who lose ≥ 10 letters from baseline to Week 12. | 9 | 0
  Participants who lose ≥ 10 letters from baseline to Week 16.: number analyzed (Participants) | 270 | 272
  Participants who lose ≥ 10 letters from baseline to Week 16. | 6 | 2
  Participants who lose ≥ 10 letters from baseline to Week 20.: number analyzed (Participants) | 263 | 269
  Participants who lose ≥ 10 letters from baseline to Week 20. | 10 | 5
  Participants who lose ≥ 10 letters from baseline to Week 24.: number analyzed (Participants) | 261 | 267
  Participants who lose ≥ 10 letters from baseline to Week 24. | 4 | 4
  Participants who lose ≥ 10 letters from baseline to Week 28.: number analyzed (Participants) | 257 | 264
  Participants who lose ≥ 10 letters from baseline to Week 28. | 9 | 8
  Participants who lose ≥ 10 letters from baseline to Week 32.: number analyzed (Participants) | 250 | 257
  Participants who lose ≥ 10 letters from baseline to Week 32. | 9 | 7
  Participants who lose ≥ 10 letters from baseline to Week 36.: number analyzed (Participants) | 252 | 259
  Participants who lose ≥ 10 letters from baseline to Week 36. | 10 | 4
  Participants who lose ≥ 10 letters from baseline to Week 40.: number analyzed (Participants) | 252 | 257
  Participants who lose ≥ 10 letters from baseline to Week 40. | 9 | 8
  Participants who lose ≥ 10 letters from baseline to Week 44.: number analyzed (Participants) | 244 | 256
  Participants who lose ≥ 10 letters from baseline to Week 44. | 6 | 9
  Participants who lose ≥ 10 letters from baseline to Week 48.: number analyzed (Participants) | 247 | 252
  Participants who lose ≥ 10 letters from baseline to Week 48. | 9 | 9
  Participants who lose ≥ 15 letters from baseline to Week 1.: number analyzed (Participants) | 280 | 275
  Participants who lose ≥ 15 letters from baseline to Week 1. | 2 | 0
  Participants who lose ≥ 15 letters from baseline to Week 4.: number analyzed (Participants) | 279 | 275
  Participants who lose ≥ 15 letters from baseline to Week 4. | 2 | 1
  Participant who lose ≥ 15 letters from baseline to Week 8.: number analyzed (Participants) | 273 | 278
  Participant who lose ≥ 15 letters from baseline to Week 8. | 1 | 0
  Participants who lose ≥ 15 letters from baseline to Week 12.: number analyzed (Participants) | 276 | 277
  Participants who lose ≥ 15 letters from baseline to Week 12. | 6 | 0
  Participants who lose ≥ 15 letters from baseline to Week 16.: number analyzed (Participants) | 270 | 272
  Participants who lose ≥ 15 letters from baseline to Week 16. | 5 | 1
  Participants who lose ≥ 15 letters from baseline to Week 20.: number analyzed (Participants) | 263 | 269
  Participants who lose ≥ 15 letters from baseline to Week 20. | 4 | 2
  Participants who lose ≥ 15 letters from baseline to Week 24.: number analyzed (Participants) | 261 | 267
  Participants who lose ≥ 15 letters from baseline to Week 24. | 1 | 2
  Participants who lose ≥ 15 letters from baseline to Week 28.: number analyzed (Participants) | 257 | 264
  Participants who lose ≥ 15 letters from baseline to Week 28. | 5 | 5
  Participants who lose ≥ 15 letters from baseline to Week 32.: number analyzed (Participants) | 250 | 257
  Participants who lose ≥ 15 letters from baseline to Week 32. | 4 | 6
  Participants who lose ≥ 15 letters from baseline to Week 36.: number analyzed (Participants) | 252 | 259
  Participants who lose ≥ 15 letters from baseline to Week 36. | 2 | 2
  Participants who lose ≥ 15 letters from baseline to Week 40.: number analyzed (Participants) | 252 | 257
  Participants who lose ≥ 15 letters from baseline to Week 40. | 3 | 5
  Participants who lose ≥ 15 letters from baseline to Week 44.: number analyzed (Participants) | 244 | 256
  Participants who lose ≥ 15 letters from baseline to Week 44. | 3 | 6
  Participants who lose ≥ 15 letters from baseline to Week 48.: number analyzed (Participants) | 247 | 252
  Participants who lose ≥ 15 letters from baseline to Week 48. | 5 | 8

6. Secondary Outcome: Percentage of Participants With BCVA Snellen Equivalent of 20/40 or Better Over Time (≥69 ETDRS Letters) for All RVO Participants.
Description: Percentage of participants with BCVA Snellen Equivalent of 20/40 or Better from Baseline to Week 48. Snellen Equivalent of 20/40 is 69 ETDRS letters. Number of participants in each treatment arm who meet specified criteria at each visit from Baseline through Week 48. Percentages are 100*n/N.
Time Frame: Day 1 - Week 48.
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | KSI-301 (Arm A) | Aflibercept (Arm B)
Number analyzed (Participants) | 284 | 284
Participants
  Snellen equivalent of 20/40 or better at Baseline. | 92 | 90
  Snellen equivalent of 20/40 or better at Week 1.: number analyzed (Participants) | 280 | 275
  Snellen equivalent of 20/40 or better at Week 1. | 168 | 153
  Snellen equivalent of 20/40 or better at Week 4.: number analyzed (Participants) | 279 | 275
  Snellen equivalent of 20/40 or better at Week 4. | 173 | 182
  Snellen equivalent of 20/40 or better at Week 8.: number analyzed (Participants) | 273 | 278
  Snellen equivalent of 20/40 or better at Week 8. | 185 | 198
  Snellen equivalent of 20/40 or better at Week 12.: number analyzed (Participants) | 276 | 277
  Snellen equivalent of 20/40 or better at Week 12. | 186 | 199
  Snellen equivalent of 20/40 or better at Week 16.: number analyzed (Participants) | 270 | 272
  Snellen equivalent of 20/40 or better at Week 16. | 200 | 209
  Snellen equivalent of 20/40 or better at Week 20.: number analyzed (Participants) | 263 | 269
  Snellen equivalent of 20/40 or better at Week 20. | 189 | 207
  Snellen equivalent of 20/40 or better at Week 24.: number analyzed (Participants) | 261 | 267
  Snellen equivalent of 20/40 or better at Week 24. | 196 | 205
  Snellen equivalent of 20/40 or better at Week 28.: number analyzed (Participants) | 257 | 264
  Snellen equivalent of 20/40 or better at Week 28. | 192 | 197
  Snellen equivalent of 20/40 or better at Week 32.: number analyzed (Participants) | 250 | 257
  Snellen equivalent of 20/40 or better at Week 32. | 182 | 190
  Snellen equivalent of 20/40 or better at Week 36.: number analyzed (Participants) | 252 | 259
  Snellen equivalent of 20/40 or better at Week 36. | 188 | 192
  Snellen equivalent of 20/40 or better at Week 40.: number analyzed (Participants) | 252 | 257
  Snellen equivalent of 20/40 or better at Week 40. | 191 | 193
  Snellen equivalent of 20/40 or better at Week 44.: number analyzed (Participants) | 244 | 256
  Snellen equivalent of 20/40 or better at Week 44. | 184 | 191
  Snellen equivalent of 20/40 or better at Week 48.: number analyzed (Participants) | 247 | 252
  Snellen equivalent of 20/40 or better at Week 48. | 182 | 190

7. Secondary Outcome: Percentage of Participants With BCVA Snellen Equivalent of 20/200 or Worse (≤ 38 ETDRS Letters) Over Time for All RVO Participants.
Description: Percentage of Participants with BCVA Snellen Equivalent of 20/200 or Worse from Baseline to Week 48. Snellen Equivalent of 20/200 is 38 ETDRS letters. Number of participants in each treatment arm who meet specified criteria at each visit from Baseline through Week 48. Percentages are 100*n/N.
Time Frame: Baseline - Week 48
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | KSI-301 (Arm A) | Aflibercept (Arm B)
Number analyzed (Participants) | 284 | 284
Participants
  Snellen Equivalent of 20/200 or Worse at Baseline | 22 | 31
  Snellen Equivalent of 20/200 or Worse at Week 1: number analyzed (Participants) | 280 | 275
  Snellen Equivalent of 20/200 or Worse at Week 1 | 9 | 12
  Snellen Equivalent of 20/200 or Worse at Week 4: number analyzed (Participants) | 279 | 275
  Snellen Equivalent of 20/200 or Worse at Week 4 | 10 | 9
  Snellen Equivalent of 20/200 or Worse at Week 8: number analyzed (Participants) | 273 | 278
  Snellen Equivalent of 20/200 or Worse at Week 8 | 6 | 5
  Snellen Equivalent of 20/200 or Worse at Week 12: number analyzed (Participants) | 276 | 277
  Snellen Equivalent of 20/200 or Worse at Week 12 | 11 | 4
  Snellen Equivalent of 20/200 or Worse at Week 16: number analyzed (Participants) | 270 | 272
  Snellen Equivalent of 20/200 or Worse at Week 16 | 7 | 7
  Snellen Equivalent of 20/200 or Worse at Week 20: number analyzed (Participants) | 263 | 269
  Snellen Equivalent of 20/200 or Worse at Week 20 | 7 | 5
  Snellen Equivalent of 20/200 or Worse at Week 24: number analyzed (Participants) | 261 | 267
  Snellen Equivalent of 20/200 or Worse at Week 24 | 2 | 4
  Snellen Equivalent of 20/200 or Worse at Week 28: number analyzed (Participants) | 257 | 264
  Snellen Equivalent of 20/200 or Worse at Week 28 | 5 | 6
  Snellen Equivalent of 20/200 or Worse at Week 32: number analyzed (Participants) | 250 | 257
  Snellen Equivalent of 20/200 or Worse at Week 32 | 3 | 5
  Snellen Equivalent of 20/200 or Worse at Week 36: number analyzed (Participants) | 252 | 259
  Snellen Equivalent of 20/200 or Worse at Week 36 | 2 | 3
  Snellen Equivalent of 20/200 or Worse at Week 40: number analyzed (Participants) | 252 | 257
  Snellen Equivalent of 20/200 or Worse at Week 40 | 2 | 7
  Snellen Equivalent of 20/200 or Worse at Week 44: number analyzed (Participants) | 244 | 256
  Snellen Equivalent of 20/200 or Worse at Week 44 | 2 | 6
  Snellen Equivalent of 20/200 or Worse at Week 48: number analyzed (Participants) | 247 | 252
  Snellen Equivalent of 20/200 or Worse at Week 48 | 5 | 8

8. Secondary Outcome: Percentage of Participants With Absence of Macular Edema (Defined as OCT CST < 325 Microns) Over Time for All RVO Participants.
Description: Macular Edema (ME) is assessed by optical coherence tomography (OCT) central subfield thickness (CST). A thickness of less than 325 microns is considered absence of ME. Proportion of participants with Absence of Macular Edema from Baseline to Week 48. Number of participants in each treatment arm who meet specified criteria at each visit from Week 1 through Week 48. Percentages are 100*n/N.
Time Frame: Baseline - Week 48
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | KSI-301 (Arm A) | Aflibercept (Arm B)
Number analyzed (Participants) | 284 | 284
Participants
  Absence of Macular Edema at Baseline | 4 | 7
  Absence of Macular Edema at Week 1: number analyzed (Participants) | 278 | 274
  Absence of Macular Edema at Week 1 | 156 | 150
  Absence of Macular Edema at Week 4: number analyzed (Participants) | 279 | 276
  Absence of Macular Edema at Week 4 | 174 | 225
  Absence of Macular Edema at Week 8: number analyzed (Participants) | 273 | 277
  Absence of Macular Edema at Week 8 | 205 | 247
  Absence of Macular Edema at Week 12: number analyzed (Participants) | 275 | 276
  Absence of Macular Edema at Week 12 | 160 | 252
  Absence of Macular Edema at Week 16: number analyzed (Participants) | 270 | 272
  Absence of Macular Edema at Week 16 | 218 | 245
  Absence of Macular Edema at Week 20: number analyzed (Participants) | 262 | 268
  Absence of Macular Edema at Week 20 | 174 | 240
  Absence of Macular Edema at Week 24: number analyzed (Participants) | 261 | 266
  Absence of Macular Edema at Week 24 | 221 | 247
  Absence of Macular Edema at Week 28: number analyzed (Participants) | 258 | 263
  Absence of Macular Edema at Week 28 | 185 | 196
  Absence of Macular Edema at Week 32: number analyzed (Participants) | 252 | 256
  Absence of Macular Edema at Week 32 | 168 | 173
  Absence of Macular Edema at Week 36: number analyzed (Participants) | 249 | 258
  Absence of Macular Edema at Week 36 | 172 | 172
  Absence of Macular Edema at Week 40: number analyzed (Participants) | 252 | 255
  Absence of Macular Edema at Week 40 | 179 | 188
  Absence of Macular Edema at Week 44: number analyzed (Participants) | 240 | 255
  Absence of Macular Edema at Week 44 | 160 | 177
  Absence of Macular Edema at Week 48: number analyzed (Participants) | 245 | 251
  Absence of Macular Edema at Week 48 | 166 | 187

9. Secondary Outcome: Mean Change in OCT Central Subfield Retinal Thickness (CST) From Baseline by Visit Over Time for All RVO Participants.
Description: Mean change in OCT central subfield retinal thickness (CST) from baseline by visit over time (up to Week 48) for all RVO participants.
Time Frame: Day 1 - Week 48
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: micrometers (um)
Arm/Group | KSI-301 (Arm A) | Aflibercept (Arm B)
Number analyzed (Participants) | 284 | 284
micrometers (um)
  Week 1: number analyzed (Participants) | 278 | 274
  Week 1 | -225.2 (152.87) | -255.9 (168.25)
  Week 4: number analyzed (Participants) | 279 | 276
  Week 4 | -230.8 (181.37) | -294.2 (195.07)
  Week 8: number analyzed (Participants) | 273 | 277
  Week 8 | -255.6 (190.40) | -310.1 (203.17)
  Week 12: number analyzed (Participants) | 275 | 276
  Week 12 | -195.8 (213.70) | -314.8 (208.68)
  Week 16: number analyzed (Participants) | 270 | 272
  Week 16 | -264.9 (204.77) | -321.0 (209.84)
  Week 20: number analyzed (Participants) | 262 | 268
  Week 20 | -218.1 (203.88) | -323.0 (209.89)
  Week 24: number analyzed (Participants) | 261 | 266
  Week 24 | -278.9 (192.68) | -326.6 (210.78)
  Week 28: number analyzed (Participants) | 258 | 263
  Week 28 | -240.4 (200.78) | -273.9 (218.56)
  Week 32: number analyzed (Participants) | 252 | 256
  Week 32 | -246.6 (200.99) | -269.7 (213.89)
  Week 36: number analyzed (Participants) | 249 | 258
  Week 36 | -243.4 (198.13) | -258.6 (213.44)
  Week 40: number analyzed (Participants) | 252 | 255
  Week 40 | -246.9 (193.79) | -274.9 (229.38)
  Week 44: number analyzed (Participants) | 240 | 255
  Week 44 | -237.5 (189.30) | -258.3 (216.49)
  Week 48: number analyzed (Participants) | 245 | 251
  Week 48 | -240.0 (203.97) | -278.8 (224.13)

10. Secondary Outcome: Mean Change in OCT Center Point Retinal Thickness (CPT) From Baseline by Visit Over Time for All RVO Participants.
Description: Mean change in OCT center point retinal thickness (CPT) from baseline by visit over time (up to Week 48) for all RVO participants.
Time Frame: Day 1 - Week 48
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: micrometers (um)
Arm/Group | KSI-301 (Arm A) | Aflibercept (Arm B)
Number analyzed (Participants) | 284 | 284
micrometers (um)
  Week 1: number analyzed (Participants) | 278 | 274
  Week 1 | -278.7 (186.23) | -320.9 (200.00)
  Week 4: number analyzed (Participants) | 279 | 276
  Week 4 | -278.5 (212.92) | -358.4 (224.51)
  Week 8: number analyzed (Participants) | 273 | 277
  Week 8 | -301.4 (220.72) | -373.9 (235.35)
  Week 12: number analyzed (Participants) | 275 | 276
  Week 12 | -230.3 (248.92) | -377.6 (239.01)
  Week 16: number analyzed (Participants) | 270 | 272
  Week 16 | -311.5 (237.01) | -381.3 (240.74)
  Week 20: number analyzed (Participants) | 262 | 268
  Week 20 | -258.1 (236.58) | -385.4 (238.61)
  Week 24: number analyzed (Participants) | 261 | 266
  Week 24 | -327.9 (223.13) | -387.5 (240.42)
  Week 28: number analyzed (Participants) | 258 | 263
  Week 28 | -280.5 (232.22) | -328.0 (249.96)
  Week 32: number analyzed (Participants) | 252 | 256
  Week 32 | -288.9 (229.6) | -322.4 (244.98)
  Week 36: number analyzed (Participants) | 249 | 258
  Week 36 | -286.8 (229.63) | -308.1 (247.22)
  Week 40: number analyzed (Participants) | 252 | 255
  Week 40 | -290.7 (220.56) | -328.7 (261.26)
  Week 44: number analyzed (Participants) | 240 | 255
  Week 44 | -281.5 (221.38) | -306.6 (252.79)
  Week 48: number analyzed (Participants) | 245 | 251
  Week 48 | -279.6 (231.43) | -331.6 (259.43)

ADVERSE EVENTS:
Time Frame: From first dose of study drug through 76 weeks. Only SAEs caused by a protocol-mandated intervention were reported from time of Informed Consent through first study intervention. After initiation of study intervention (Day 1) through final safety follow-up visit, all AE and SAE information were collected.
Groups:
- KSI-301 (Arm A): Intravitreal injection of KSI-301 (5 mg) at Day 1, Week 4, and once every 8 weeks through Week 20 followed by an individualized dosing regimen of Intravitreal injection of KSI-301 (5 mg) from Week 24 to Week 44.
  KSI-301: Intravitreal Injection
  Sham Procedure: The sham is a procedure that mimics an intravitreal injection. It involves pressing the blunt end of an empty syringe (without a needle) against the anesthetized eye. It will be administered to participants in both treatments arms at applicable visits to maintain masking.
- Aflibercept (Arm B): Intravitreal injection of aflibercept (2 mg) once every 4 weeks through Week 20 followed by an individualized dosing regimen of Intravitreal injection of Aflibercept (2 mg) once every 4 weeks from Week 24 to Week 44.
  Aflibercept: Intravitreal Injection
  Sham Procedure: The sham is a procedure that mimics an intravitreal injection. It involves pressing the blunt end of an empty syringe (without a needle) against the anesthetized eye. It will be administered to participants in both treatments arms at applicable visits to maintain masking.
- KSI-301 5mg Extension Phase: In the Extension Phase, participants randomized to KSI-301 (5 mg) in the Primary Study will continue to receive KSI-301 (5 mg) based on protocol-defined disease activity criteria.
  In the Extension Phase, participants randomized to aflibercept in the Primary Study will cross over to treatment with KSI-301 (5 mg). They will receive their first dose of KSI-301 (5 mg) at Week 48 and will receive additional treatment with KSI-301 (5 mg) based on protocol-defined disease activity criteria.
Arm/Group | KSI-301 (Arm A) | Aflibercept (Arm B) | KSI-301 5mg Extension Phase
All-Cause Mortality (participants affected / at risk) | 3/284 | 1/284 | 2/444
Serious Adverse Events (participants affected / at risk) | 36/284 | 23/284 | 18/444
Other Adverse Events (participants affected / at risk) | 73/284 | 66/284 | 53/444
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | KSI-301 (Arm A) (N=284) | Aflibercept (Arm B) (N=284) | KSI-301 5mg Extension Phase (N=444)
Atrial fibrillation (Cardiac disorders) | 2 (3) | 2 (2) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrioventricular block (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (3) | 1 (1) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Furuncle (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Vestibular neuronitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Epididymitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Orchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Retinal detachment - Fellow eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Glaucoma - Study eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Lens dislocation - Study eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Rhegmatogenous retinal detachment - Study eye (Eye disorders) | 1 (2) | 0 (0) | 0 (0)
Vitritis - Study eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Retinal vein occlusion - Study eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fractured sacrum (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Waldenstrom's macroglobulinaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Myelopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (2) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Arteriosclerosis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Giant cell arteritis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Intraocular pressure increased - Study eye (Investigations) | 1 (1) | 0 (0) | 0 (0)
Device malfunction (Product Issues) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Volvulus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 2 (2) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Dementia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Lacunar infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Nerve compression (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Bronchial neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Sarcomatoid carcinoma of the lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Essential hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Shock (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Retinal detachment - Study Eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | KSI-301 (Arm A) (N=284) | Aflibercept (Arm B) (N=284) | KSI-301 5mg Extension Phase (N=444)
Conjunctival haemorrhage - Study eye (Eye disorders) | 24 (27) | 22 (24) | 8 (8)
COVID-19 (Infections and infestations) | 30 (30) | 23 (23) | 32 (33)
Hypertension (Vascular disorders) | 30 (31) | 26 (28) | 13 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2021-06-02): https://cdn.clinicaltrials.gov/large-docs/19/NCT04592419/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-22): https://cdn.clinicaltrials.gov/large-docs/19/NCT04592419/SAP_001.pdf